CLINICAL TRIAL: NCT00880919
Title: Seroquel XR for the Management of Borderline Personality Disorder (BPD)
Brief Title: Seroquel Extended Release (XR) for the Management of Borderline Personality Disorder (BPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: AstraZeneca (Industry); University of Iowa (Other); Mclean Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0709M16844; IRUSQUET0454 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; BPD; Seroquel; Seroquel XR; quetiapine; quetiapine extended-release
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Seroquel XR 150mg oral tablets taken daily for 8 weeks.
  Interventions: Drug: quetiapine extended-release
- 2 (Active Comparator): Seroquel XR 300mg oral tablets taken daily for 8 weeks.
  Interventions: Drug: quetiapine extended-release
- 3 (Placebo Comparator): Equivalent number of placebo oral tablets taken daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: quetiapine extended-release — Seroquel XR 150mg/day vs Seroquel XR 300mg/day vs Placebo
  Other Names: Seroquel XR
  Arms: 1; 2
Drug: Placebo — Seroquel XR 150mg/day vs Seroquel XR 300mg/day vs Placebo
  Other Names: quetiapine extended-release
  Arms: 3

SUMMARY:
The Primary objective of this study is to evaluate Seroquel XR in the treatment of borderline personality disorder (BPD). As in many initial randomized control trials, the study will be of relatively short duration - 8 weeks - to assess effectiveness and safety while maximizing retention. The specific aim is to determine if Seroquel XR is superior to placebo. The primary outcome measure will be a statistically significant difference between Seroquel XR compared to placebo on the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD), an objective rating scale that addresses the severity of Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) symptoms of the illness. As there is the recent development of an extended release form of Seroquel (Seroquel XR) (Schulz et al. 2007), the new compound may offer several advantages in this study. Therefore, the hypothesis of this study is that both doses of Seroquel XR (see below) will be superior to placebo in an 8-week randomized trial as assessed by the ZAN-BPD.

To achieve the Primary Objective of this study, two doses of Seroquel XR will be tested - 150 mg/d and 300 mg/d. Thus, the study will be able to assess the effect of Seroquel XR compared to placebo and to explore a dose effect.

DETAILED DESCRIPTION:
The secondary objectives in this study are aimed at answering further questions regarding symptom assessments, dosing strategies, and safety. The specific secondary objectives are listed below:

1. Response rate: In previous studies using the ZAN-BPD, response was defined as a 50% reduction of ZAN-BPD scores. Response rates will be compared between Seroquel XR and placebo.
2. Other Symptom Measures: Over the last twenty years, other rating scales of a general nature have been used to assess BPD patients in clinical trials. To fully assess the patients as they progress through the study, the following scales will be administered: Symptom Checklist 90 - Revised (SCL-90 R), Montgomery Asberg Depression Rating Scale (MADRS), Barratt Impulsivity Scale (BIS), Schedule for Interviewing Borderlines (SIB), Overt Aggression Scale - Modified (OAS-M), Young Mania Rating Scale (YMRS), the Borderline Evaluation of Severity over Time (BEST), and the Global Assessment of Function (GAF).
3. Side-Effects: To be able to report the safety of Seroquel XR for BPD, a combination of objective and subjective measures will be employed. Objectively, weight, height (and Body Mass Index (BMI)), prolactin, glucose, cholesterol and triglycerides will be assessed at baseline and endpoint. Objective ratings of movement side effects will be performed using Simpson Angus Scale (SAS) (Simpson and Angus 1970), Barnes Akathisia Scale (BAS) (Barnes 1989), and Abnormal Involuntary Movement Scale (AIMS) (Guy 1976), and at baseline and endpoint. Regarding possible side effects reported by patients, their reports of headache, somnolence, and other experiences will be tabulated.

Secondary objective data will be analyzed as continuous variable data over the time of the study or, when appropriate, comparisons of baseline to endpoint will be made.

ELIGIBILITY:
Inclusion Criteria:

* Consent
* A diagnosis of borderline personality disorder (301.83)
* All subjects will have a ZAN-BPD greater or equal to 9 at randomization.
* Males and females aged 18-45 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Pregnancy or lactation
* Any DSM-IV Axis I disorder not defined in the inclusion criteria. The patients with BPD may not have bipolar I disorder, schizophrenia, schizoaffective disorder, delirium, or dementia. Neither may they have current DSM-IV substance dependence.
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine, and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension, congestive heart failure) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study.
* Participation in another drug trial within 4 weeks prior enrollment into this study or longer in accordance with local requirements
* Unstable Diabetes Mellitus
* An absolute neutrophil count (ANC) of 1.5 x 109 per liter
* Past history of lack of response to an atypical antipsychotic medication or substantial previous side effects will be cause for exclusion.
* Any medical illness that would interfere with conduct of the study will be cause for exclusion.
* Pregnant or lactating women and women of childbearing potential not using medically accepted means of contraception.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2008-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Charles Schulz, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Iowa, Department of Psychiatry, Iowa City, Iowa
  - McLean Hospital, Harvard Medical School, Department of Psychiatry, Belmont, Massachusetts
  - University of Minnesota Medical Center, Fairview Riverside, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind, placebo-controlled, dose comparison trial was conducted at three outpatient treatment centers from January 2010 to March 2013.
Pre-assignment Details: Ninety-five persons with Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) borderline personality disorder (BPD) were randomly assigned to quetiapine XR 150 mg/day (n=33), quetiapine XR 300 mg/day (n=33), or placebo (n=29).
Groups:
- Quetiapine XR 150 mg/Day (n=33),: Seroquel XR 150mg oral tablets taken daily for 8 weeks.
- Quetiapine XR 300 mg/Day (n=33),: Seroquel XR 300mg oral tablets taken daily for 8 weeks.
- Placebo (n=29).: Equivalent number of placebo oral tablets taken daily for 8 weeks.
Period: Overall Study
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Started | 33 | 33 | 29
Completed | 18 | 19 | 23
Not Completed | 15 | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29). | Total
Number analyzed (Participants) | 33 | 33 | 29 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 29 | 95
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (8.0) | 30.2 (8.1) | 20.1 (8.8) | 29.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 19 | 67
  Male | 8 | 10 | 10 | 28
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 29 | 95

OUTCOME MEASURES:

1. Primary Outcome: Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD)
Description: This is an assessment of change in DSM-IV borderline psychopathology. Consisting of nine criteria rated on a five-point anchored rating scale of 0 to 4, yielding a total score of 0 to 36. 0 being the best and 4 meaning the worse.
Time Frame: baseline, weekly until week 8
Population: All subjects randomly assigned to a treatment group were included in the intent-to-treat analyses of baseline demographic and clinical characteristics. The efficacy analyses were limited to subjects with at least one post-randomization observation to guarantee measurement of change.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -1.22 (0.15) | -0.99 (0.16) | -0.75 (0.15)
Statistical Analysis 1: Comparison: Quetiapine XR 150 mg/Day (n=33), vs Quetiapine XR 300 mg/Day (n=33), vs Placebo (n=29); Mean changes were calculated using each groups linear and quadratic effects; Test type: Superiority or Other; p = .015, ANOVA

2. Primary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: Nine criteria rated on a six-point anchored rating scale of 0 to 6, yielding a total score of 0 to 60. O is the least and 6 is the highest
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Quetiapine XR 150 mg/Day (n=33): Seroquel XR 150mg oral tablets taken daily for 8 weeks.
  quetiapine extended-release: Seroquel XR 150mg/day vs Seroquel XR 300mg/day vs Placebo
- Quetiapine XR 300 mg/Day (n=33): Seroquel XR 300mg oral tablets taken daily for 8 weeks.
  quetiapine extended-release: Seroquel XR 150mg/day vs Seroquel XR 300mg/day vs Placebo
- Placebo (n=29): Equivalent number of placebo oral tablets taken daily for 8 weeks.
  Placebo: Seroquel XR 150mg/day vs Seroquel XR 300mg/day vs Placebo
Arm/Group | Quetiapine XR 150 mg/Day (n=33) | Quetiapine XR 300 mg/Day (n=33) | Placebo (n=29)
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -0.85 (0.19) | -1.05 (0.19) | -0.59 (0.18)

3. Primary Outcome: Borderline Evaluation of Severity Over Time (BEST)
Description: Scale including 15 items and three subscales. All items are rated on a Likert-like scale. A correction factor of 15 is added to yield the final score which can range from 12 (best) to 72 (worst).
Time Frame: Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -2.10 (0.32) | -1.97 (0.33) | -0.91 (0.31)

4. Primary Outcome: Overt Aggression Scale - Modified (OAS-M)
Description: Four part behavior rating scale designed to measure four types of aggressive behavior as witnessed in the past week. Each section consists of five questions. Total scores on the MOAS range from 0-40. 0 is the best and 40 is the worst of symptoms Reduction in scores shows a change of symptoms.
Time Frame: Change from Baseline Overt Aggression Scale - Modified to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -1.92 (0.42) | -1.82 (0.43) | -0.37 (0.43)

5. Primary Outcome: Global Assessment of Functioning Scale (GAF)
Description: Numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults. 100 is the highest level of functioning. O is the least functional
Time Frame: Change in Global Assessment of Functioning from Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | 1.05 (0.20) | 1.04 (0.21) | 0.62 (0.19)

6. Primary Outcome: Barratt Impulsiveness Scale (BIS)
Description: 30-item self-report questionnaire, that is scored to yield a total score, three second-order factors, and six first-order factors. patients rate the questions 1-4 1 being the least and 4 being the most.
Time Frame: Change in Impulsiveness from Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -0.73 (0.27) | -0.83 (0.27) | -.59 (0.26)

7. Primary Outcome: Symptom Checklist -90-Revised (SCL-90-R)
Description: 90 items measured on a Likert scale via self-report. Scale is 0-5 stating 0= strongly disagree and 5 is Strongly agree Measures psychological problems and symptoms
Time Frame: Change in psychological problems and symptoms from Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -0.11 (0.02) | -0.12 (0.02) | -0.07 (0.02)

8. Primary Outcome: Young Mania Rating Scale (YMS)
Description: Eleven-item multiple choice diagnostic questionnaire, yielding total scores of 0-60. 0-4 rating 0-being least likely and 4 being most likely This scale assess manic symptoms
Time Frame: Change in manic symptoms from Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -0.26 (0.06) | -0.30 (0.06) | 0.11 (0.06)

9. Primary Outcome: Sheehan Disability Scale (SDS)
Description: Three self-rated items, on a scale of 0-10. 0 is unimpaired 10 is highly impaired This measures functional impairment
Time Frame: Change in functional impairment from Baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Number analyzed (Participants) | 33 | 33 | 29
units on a scale | -0.85 (0.19) | -1.11 (0.20) | 0.58 (0.18)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Quetiapine XR 150 mg/Day (n=33), | Quetiapine XR 300 mg/Day (n=33), | Placebo (n=29).
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 29/33 | 30/33 | 19/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine XR 150 mg/Day (n=33), (N=33) | Quetiapine XR 300 mg/Day (n=33), (N=33) | Placebo (n=29). (N=29)
Sedation (Nervous system disorders) | 29 (29) | 30 (30) | 19 (19)
Change in appetite (Metabolism and nutrition disorders) | 9 (9) | 12 (12) | 4 (4)
Dry mouth (General disorders) | 9 (9) | 14 (14) | 1 (1)
Headache (General disorders) | 7 (7) | 10 (10) | 6 (6)
Bodily pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) | 5 (5)
Hypersomnia (General disorders) | 5 (5) | 8 (8) | 2 (2)
Dizziness (General disorders) | 5 (5) | 7 (7) | 1 (1)
Forgetfulness or confusion (Nervous system disorders) | 5 (5) | 7 (7) | 1 (1)
Nausea or vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No